CLINICAL TRIAL: NCT06654492
Title: Retrospective Study of Small Window Lateral Maxillary Sinus Floor Elevation Surgery
Brief Title: The Systematic Evaluation of the Surgery, Using the Ratio of the Window Area to the Volume of Bone Graft Material
Status: Completed | Type: Observational
Sponsor: Kunming Medical University (Other)
Responsible Party: Principal Investigator, Fangyu Yao, Graduate student, Kunming Medical University
Other Study IDs: KYKQ2024MEC0050
Record Dates: First submitted 2024-10-17; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Maxillary Sinus Floor Elevation
Keywords: LW-MSFE

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The cylindrical bone tissue extracted from the implant site half a year after the small lateral window maxillary sinus floor elevation surgery has a diameter of approximately 3 millimeters and a height of 5 millimeters. This bone tissue is used for Micro-CT scanning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: The dimension of the window for lateral window maxillary sinus elevation surgery — The window size for a single implant site should not exceed 25 square millimeters, while the window size for consecutive multiple implant sites should not exceed 40 square millimeters.

SUMMARY:
Objective: To conduct a systematic mid-to-long-term efficacy evaluation of the small window lateral maxillary sinus floor elevation surgery, using the ratio of the window area to the volume of bone graft material as an innovative evaluation metric; to provide clinical evidence for the treatment and assessment of maxillary sinus elevation surgery. Research Content and Methods: The study included all patients who underwent lateral wall small window surgery performed by Dr. Xie Liangkun from 2017 to 2024 in Affiliated Stomatology Hospital of Kunming Medical University. Seventy-seven patients underwent cone-beam computed tomography (CBCT) at each stage before grafting, before the surgery,immediately after the surgery, 6 months postoperatively, and after tooth placement. The CBCT data were imported into Mimics software to measure the volume of bone graft material at different periods (b value), and The photos which recording window size during surgery were imported into ImageJ software to measure the window area (a value). CBCT was also used to measure the distance from the window to the sinus floor, the thickness of the lateral wall bone plate, and the thickness of the Schneiderian membrane as secondary measurement indicators. The ratio of a/b was statistically analyzed for correlation with various secondary indicators, and conclusions were drawn. Bone cores taken 6 months after grafting (before implant placement) were subjected to Micro-CT scanning and histological analysis to evaluate the bone formation effects.

DETAILED DESCRIPTION:
Research significance:The first part is the elevation of maxillary sinus floor through minimally invasive window side wall small window. Through retrospective study of implant retention rate, complications, patient subjective perception, anatomical factors and other indicators, it is used to comprehensively evaluate the clinical efficacy of this surgical procedure. In the second part, representative bone columns are taken for Micro CT scanning to evaluate the osseointegration from a histological perspective. Mimics software performs three-dimensional scanning of the transplant area, and the ratio of the window area to the volume of the transplant part is used as the main measurement index to demonstrate that minimally invasive window opening can achieve ideal bone grafting effects. Further verify the success or failure of minimally invasive side wall fenestration surgery. At present, relevant studies use this ratio as the main research data, and there is no use of 3D scanning to study changes in bone transplant areas. There are also few studies evaluating the binding of bone tissue using Micro CT, and most of them use CBCT 2D measurement data for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older;
2. Missing posterior maxillary teeth;
3. The missing tooth area has been edentulous for at least 3 months;
4. No acute severe maxillary sinus inflammation, and no tumor or other space-occupying lesions within the maxillary sinus;
5. The residual bone height (RBH) in the missing tooth area is less than 4mm;
6. Sufficient alveolar bone width in the missing tooth area to ensure implant placement;
7. Signed an informed consent form and can return for follow-up visits as scheduled.

Exclusion Criteria:

1. Patients with systemic diseases not suitable for implantation: such as uncontrolled hypertension, diabetes, cardiovascular and cerebrovascular diseases, bone metabolic diseases, head and face radiotherapy, etc.;
2. Uncontrolled periodontitis or mucosal disease patients;
3. Patients with bruxism;
4. Patients who have undergone implant placement or artificial bone material implantation in the missing tooth area;
5. Patients with mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collected all patients who underwent small lateral window maxillary sinus elevation surgery performed by Dr. Xie Liangkun from 2017 to 2024.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
The window area of the lateral wall maxillary sinus floor elevation surgery | immediately after surgery
  intraoperative window photos were imported into ImageJ software to measure the window area (a value)

SECONDARY OUTCOMES:
the volume of bone graft material | before implant surgery, immediately after surgery，6 months after surgery
  Import the CBCT scans from immediately after surgery, half a year postoperatively, and after tooth placement into the Mimics software to measure the volume

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Xie, Principal Investigator — Kunming Medical University
Locations (1):
- Kunming Medical University, Kunming, Yunan, China

IPD SHARING:
Plan to Share IPD: Undecided